CLINICAL TRIAL: NCT03425318
Title: Continuous Negative Abdominal Pressure in ARDS (CNAP in ARDS)
Acronym: CNAP in ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head Respiratory Medicine, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000060365
Record Dates: First submitted 2018-01-29; First posted 2018-02-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients with ARDS will be placed inside of a Continuous Negative Abdominal Pressure Device. Negative pressure will be applied to the abdomen as an adjunct to positive pressure ventilation
  Interventions: Device: CNAP

INTERVENTIONS:
Device: CNAP — Application of CNAP in patients with ARDS

SUMMARY:
The aim is to test a device for applying continuous negative abdominal pressure in patients with ARDS

DETAILED DESCRIPTION:
Adult respiratory distress syndrome (ARDS) is a serious pulmonary disease affecting adults and children. It has a high mortality and there is no specific therapy. The mortality is high (approx. 40% in severe cases) and this has not changed in the last 20 years.

Mechanical ventilation is the mainstay of management, and this assists the patient by increasing oxygenation and removal of carbon dioxide. Despite optimizing tidal volume, driving pressure and positive end-expiratory pressure (PEEP), patients with ARDS develop large areas of atelectasis and poor oxygenation. There are few additional ventilator approaches that have proven to be useful in preventing this type of injury.

A major aim of ventilator support is recruitment of atelectatic (i.e. de-airated) lung, but while this is supported by excellent rational and laboratory data, the conventional clinical approaches have not been associated with a demonstrable improvement in patient outcome. Most atelectasis in ARDS occurs in the dorsal (dependant, lower-most) lung regions, and these are near the diaphragm.

The main ways to recruit lung are to increase the airway distending pressure (but this over-expands and damages the already-aerated lung regions); or, to turn the patient into the prone position (but clinicians are reluctant to utilize this approach - despite evidence that it may increase survival).

Continuous Negative Abdominal Pressure (CNAP) aims to selectively recruit basal atelectatic areas of lung, while enabling the patient to remain in the supine (usual) position.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≧ 18 years old
2. Patients with moderate to severe ARDS as per the Berlin definition (PaO2/FiO2 ≤200mmHg)
3. Patients with absence of any significant cardiopulmonary disease

Exclusion Criteria:

1. Contraindication to CNAP

   a. open abdominal wounds or drainage tubes; b. Acute brain Injury with intracranial pressure >30 mm Hg or cerebral perfusion pressure <60 mmHg; c. Decompensated heart insufficiency or acute coronary syndrome; d. Major hemodynamic instability: Mean arterial pressure lower than 60 mm Hg despite adequate fluid resuscitation and two vasopressors or increase of vasopressor dose by 30% in the next 6 hours; f. Unstable spine, femur, or pelvic fractures; g. Pregnancy; h. Pneumothorax;
2. Contraindication to EIT electrode placement: Burns, chest wall bandaging limiting electrode placement
3. Severe liver insufficiency (Child-Pugh score > 7) or fulminant hepatic failure
4. Major respiratory acidosis or PaCO2 > 60 mmHg
5. Severe COPD (according to the GOLD criteria defined as severe = FEV1: 30-50% or very severe = FEV1 < 30%)
6. Clinical judgement of the attending physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hypotension (SAFETY) | 30 min
  Reduction in mean arterial pressure to less than 60 mmHg or by 15%
Oxygen Saturation (SAFETY | 30 min
  Reduction in oxygen saturation (SpO2) by 5% or more
Oxygenation (SAFETY) | 30 min
  Reduction in P-to-F ratio (PaO2/FiO2) by >20%

SECONDARY OUTCOMES:
Oxygenation (EFFICACY) | 30 min
  Increase in PaO2/FiO2 by >20%

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03425318/Prot_SAP_000.pdf